CLINICAL TRIAL: NCT01854476
Title: A Double-bline Safety and Efficacy Study Comparing Pad-gauze With Tranexamic Acid (Hemostopan™) to a Regular Pad-gauze in Controlling Bleeding in Patients on Hemodialysis.
Brief Title: Safety and Efficacy Study Comparing Pad-gauze With Anti-fibrinolytic Agent Hemostopan™) to a Regular Pad-gauze
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sion Microtec Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SionM1
Record Dates: First submitted 2013-05-12; First posted 2013-05-15 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Bleeding; Coagulopathy
Keywords: Hemodialysis; Bleeding; Hemostatic dressing; Tranexamic Acid
MeSH Terms: conditions — Hemorrhage; Hemostatic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic acid (Experimental): pad-gauze with tranexamic acid (Hemostopan™)
  Interventions: Device: pad-gauze with tranexamic acid (Hemostopan™)
- Pad gauze (Placebo Comparator): Pad gauze with no tranexamic acid

INTERVENTIONS:
Device: pad-gauze with tranexamic acid (Hemostopan™) — The use of pad-gauze containing tranexamic acid (Hemostopan™)
  Arms: Tranexamic acid

SUMMARY:
Patients on chronic treatment with hemodialysis have an arterio-venous fistula which enable the insertion of two large gauge needles. At the end of dialysis the needles are extracted and continuous pressure is needed to stop the bleeding. Time to bleeding cessation is different between patients and may be up to 20 minutes. Acquired coagulopathy in patients on chronic hemodylasis is a well known entity. The coagulopathy is multi-factorial including uremic thrombocytopathia, the presence of anemia, the use of anti-platelets and/or anti-coagulation drugs and the regular use of heparin during dialysis. Tranexamic acid (Hexakapron) is an anti-fibrinolytic drug that has a proven efficacy in reducing blood loss at different clinical settings. The drug may be given systemically (PO/IV) or applied locally on the site of injury.

The aim of the study is to assess the efficacy and safety of a pad gauze dressing containing tranexamic acid.

Study design:

A Double-blind study comparing pad-gauze with tranexamic acid (Hemostopan™) to a regular pad-gauze. The type of dressing for each dialysis session will be decided in a random manner. In each dialysis session only one type of dressing will be used for both insertion points.

Protocol for applying the dressing:

Following the needle extraction either dressing "A" or "B" will applied with slight pressure for 2 minutes. If bleeding stops it will be the end of session.

If bleeding persists than another dressing of the same kind is applied with slight pressure for 4 minutes. If bleeding stops it will be the end of session.

If bleeding persists than another dressing of the same kind is applied with slight pressure for 6 minutes. If bleeding stops it will be the end of session.

If bleeding persists than it will be consider a failure and a regular measures will be used until bleeding stops.

Each session will be documented in the patient's case report file (CRF). The primary end point of the study: Time to bleeding cessation

DETAILED DESCRIPTION:
A Double-blind safety and efficacy study comparing pad-gauze with tranexamic acid (Hemostopan™) to a regular pad-gauze in controlling bleeding in patients on hemodialysis.

Background:

Patients with end-stage renal disease are on chronic treatment with hemodialysis. Most patients have and arterio-venous fistula which enable the insertion of two large gauge needles. At the end of dialysis the needles are extracted and continuous pressure is needed to stop the bleeding. Time to hemostasis is different between patients and may be up to 20 minutes for each insertion point. Acquired coagulopathy in patients on chronic hemodylasis is a well known entity which have an important impact on time to hemostasis. The coagulopathy is multi-factorial composed including uremic thrombocytopathia, the presence of anemia, the use of anti-platelets and / or anti-coagulation drugs and the regular use of heparin during the dialysis process. Tranexamic acid (Hexakapron) is an anti-fibrinolytic drug that has a proven efficacy in reducing blood loss at different clinical settings. The drug may be given systemically (PO / IV) or applied locally on the site of injury.

The aim of the study To study the efficacy and safety of a pad gauze dressing containing tranexamic acid.

Inclusion criteria:

Patients that requires at least 10 minutes for hemostasis will be considered candidates for the study. Among those, only patient over 18 years of age that will sign an informed consent will be recruited.

Exclusion criteria:

Patients with HIV, HCV or HBV chronic infection. Known hypersensitivity to polydine.

Study design:

A Double-blind study comparing pad-gauze with tranexamic acid (Hemostopan™) to a regular pad-gauze. The type of dressing for each dialysis session will be decided in a random manner. In each dialysis session only one type of dressing will be used for both insertion points. The dressing are identical in their appearance and are marked as dressing "A" or dressing "B". All of the participants including - patients, physician, nurses and study coordinator will be blinded to the treatments. In ta course of the study each dressing will be applied 10 times in a given patient so in practical each patient will be his own control.

Protocol for applying the dressing:

Following the needle extraction either dressing "A" or "B" will applied with slight pressure for 2 minutes. If bleeding stops it will be the end of session.

If bleeding persists than another dressing of the same kind is applied with slight pressure for 4 minutes. If bleeding stops it will be the end of session.

If bleeding persists than another dressing of the same kind is applied with slight pressure for 6 minutes. If bleeding stops it will be the end of session.

If bleeding persists than it will be consider a failure and a regular measures will be used until bleeding stops.

Each session will be documented in the patient's case report file (CRF).

The primary end point of the study:

Time to hemostasis

ELIGIBILITY:
Inclusion Criteria:

* Patients that require at least 10 minutes for hemostasis
* Patient over 18 years of age that are capable of signing an informed consent

Exclusion Criteria:

* Patients with HIV, HCV or HBV chronic infection
* Known hypersensitivity to polydine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Time to hemostasis | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mudi Misgav, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- The dialysis unite at the Sheba Medical center, Ramat Gan, Israel, Israel

REFERENCES:
- [Background] 1.Remuzzi G, Livio M, Marchiaro G, Mecca G, de Gaetano G.Bleeding in renal failure: altered platelet function in chronic uraemia only partially corrected by haemodialysis. Nephron. 1978;22(4-6):347-53. 2.Akizawa T, Kinugasa E, Kitaoka T, Koshikawa S. Effects of recombinant human erythropoietin and correction of anemia on platelet function in hemodialysis patients. Nephron 1991;58:400-6. 3.Mezzano D, Panes O, Muñoz B, Pais E, Tagle R, González F, Mezzano S, Barriga F, Pereira J.Tranexamic acid inhibits fibrinolysis, shortens the bleeding time and improves platelet function in patients with chronic renal failure. ThrombHaemost. 1999 Oct;82(4):1250-4. 4.Saran R, Pisoni RL, Weitzel WF. Epidemiology of vascular access for hemodialysis and related practice patterns. ContribNephrol 2004; 142: 14-28. 5.Wu CC, Ho WM, Cheng SB, Yeh DC, Wen MC, Liu TJ, P'eng FK. Perioperative parenteral tranexamic acid in liver tumor resection: a prospective randomized trial toward a